CLINICAL TRIAL: NCT02431910
Title: Immediate and Delayed Effects of Kinesio Taping on the Neuromuscular Performance, Balance and Lower Limb Function of Healthy Subjects: Randomized Clinical Trial
Brief Title: Immediate and Delayed Effects of Kinesio Taping on the Neuromuscular Performance
Acronym: IDEKTNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Jamilson Simões Brasileiro, Professor of Physiotherapy, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 752.302
Record Dates: First submitted 2015-04-09; First posted 2015-05-01 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Neuromuscular Performance, Balance and Function
Keywords: Electromyography; Baropodometry; Torque

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (No Intervention): The control group remains at rest for 10 minutes, which is not applied KT in the RF, VL and VM muscles. The volunteers of this group perform all evaluation without the application of KT
- Placebo group (Placebo Comparator): The Kinesio Taping (KT) is applied on the vastus lateralis (VL), vastus medialis (VM) and rectus femoris (RF) muscles longitudinally from proximal to the distal. For the RF proximal anchor is applied 5cm below the anterior superior iliac spine and the distal anchor the upper edge of the patella. VL in the proximal and distal anchor will be fixed in greater trochanter of the femur and the lateral edge of the patella. As for the VM muscle proximal anchor will be applied to the middle third from the medial region of the thigh and the distal anchor on the medial edge of the patella. The anchors are applied with 0% tension and therapy area will follow on the belly of the muscles with a 0%.
  Interventions: Other: placebo Functional elastic tape
- Kinesio Taping group (Experimental): The Kinesio Taping (KT) is applied on the vastus lateralis (VL), vastus medialis (VM) and rectus femoris (RF) muscles longitudinally from proximal to the distal. For the RF proximal anchor is applied 5cm below the anterior superior iliac spine and the distal anchor the upper edge of the patella. VL in the proximal and distal anchor will be fixed in greater trochanter of the femur and the lateral edge of the patella. As for the VM muscle proximal anchor will be applied to the middle third from the medial region of the thigh and the distal anchor on the medial edge of the patella. The anchors are applied with 0% tension and therapy area will follow on the belly of the muscles with a 50%. This application will be held with subjects standing on one foot, with the hip of the non-dominant limb at 0º and knee flexed at 90º.
  Interventions: Other: Functional elastic tape

INTERVENTIONS:
Other: Functional elastic tape — application of KT with tension in the vastos medialis, rectus femoris and vastus lateralis muscles
  Other Names: Kinesio Taping
  Arms: Kinesio Taping group
Other: placebo Functional elastic tape — application of KT without tension in the vastos medialis, rectus femoris and vastus lateralis muscles
  Other Names: placebo Kinesio Taping
  Arms: Placebo group

SUMMARY:
The purpose of this study is analyze the immediate and late effects of the application of KT in neuromuscular performance of the quadriceps in postural balance and function of the lower limb of healthy subjects.

DETAILED DESCRIPTION:
Sixty volunteers, females will be recruited and randomly divided into 3 groups with 20 members each: control group (CG) - 10 minutes at rest; placebo group (PG) - Kinesio Taping (KT) without application of tension in the vastus lateralis (VL), vastus (VM) and rectus femoris (RF); and Kinesio Taping group (KTG) - application of KT with tension in VL, VM and RF. All volunteers will be evaluated for their distance from the single and triple hop test, postural balance (baropodometry), the joint position sense (JPS), the knee extensor torque (concentric and eccentric assessment at 60 °/s) and electromyographic activity of the VL muscle in five distinct stages: the first before the intervention (AV1), the second immediately after (AV2) and the following three 24h (AV3), 48 (AV4) after the intervention protocol. Soon after the AV4, KT will be removed after 24 hours and take place the last review (AV5).

ELIGIBILITY:
Inclusion Criteria:

* Be recreationally active, with no history of osteomyoarticular lesion or surgery in the lower limbs in the previous six months, non-corrected neurological, vestibular, visual and/or hearing impairments, in addition to displaying no allergy to adhesive material.

Exclusion Criteria:

* Individuals experiencing pain during collection procedures or who do not perform exercises as instructed by the researchers would be excluded.

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Muscle Performance measured through isokinetic dynamometry | baseline, one minute after the intervention protocol, 24 hours, 48 hours and 72 hours after the intervention protocol.
  Change from baseline in muscle performance at 72 hours.Immediate and Delayed Effects of Kinesio Taping in the muscle performance will be measured through isokinetic dynamometry and the variables analyzed will be peak torque normalized for body weight, mean power, total work and time to peak torque.

SECONDARY OUTCOMES:
Balance measured through baropodometry | baseline, one minute after the intervention protocol, 24 hours, 48 hours and 72 hours after the intervention protocol.
  Change from baseline in balance at 72 hours. Immediate and Delayed Effects of Kinesio Taping in balance will be Measured by baropodometry
Lower limb function | baseline, one minute after the intervention protocol, 24 hours, 48 hours and 72 hours after the intervention protocol.
  Change from baseline in lower limb function at 72 hours. Immediate and Delayed Effects of Kinesio Taping will be measure through distance of the single and triple hop test.
Proprioception measured through joint position sense in the isokinetic dynamometer | baseline, one minute after the intervention protocol, 24 hours, 48 hours and 72 hours after the intervention protocol.
  Change from baseline in proprioception at 72 hours. Immediate and Delayed Effects of Kinesio Taping in the proprioception will be measured through joint position sense
Muscle activation measured through surface electromyography | baseline, one minute after the intervention protocol, 24 hours, 48 hours and 72 hours after the intervention protocol.
  Change from baseline in muscle activation at 72 hours. Immediate and Delayed Effects of Kinesio Taping in Muscle activation will be Measured by surface electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Jamilson S Brasileiro, PhD, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Universidade Federal do Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil